CLINICAL TRIAL: NCT01327547
Title: A Multicenter, Randomized, Blinded, Placebo-controlled Study To Evaluate The Safety Of Maraviroc In Combination With Other Antiretroviral Agents In Hiv-1-infected Subjects Co-infected With Hepatitis C And/or Hepatitis B Virus
Brief Title: A Study Of Maraviroc In HIV Co-Infected Subjects With Hepatitis C And/Or Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4001098; 2010-021994-35 (EudraCT Number)
Record Dates: First submitted 2011-03-22; First posted 2011-04-01 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: HIV Coinfection
Keywords: HIV coinfection; maraviroc; CCR5 blocker; entry inhibitor; liver disease; viral hepatitis
MeSH Terms: conditions — HIV Infections; Liver Diseases | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1.0 (Experimental)
  Interventions: Drug: Maraviroc
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maraviroc — 150mg, 300mg or 600mg twice daily x 144 weeks; dosing dependent on components of the current suppressive anti-HIV therapy
  Other Names: Selzentry, Celsentri
  Arms: 1.0
Drug: Placebo — 150mg, 300mg or 600mg twice daily x 144 weeks; dosing dependent on components of the current suppressive anti-HIV therapy
  Arms: 2

SUMMARY:
To describe liver enzyme elevations in patients who are coinfected with HIV and either Hepatitis C (HCV) and/or Hepatitis B (HBV) receiving maraviroc or placebo in combination with their current suppressive anti-HIV drug therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV coinfected with HCV and/or HBV.
* Undetectable HIV-1 RNA for at least 3 months prior to the screening visit
* Treatment with current antiretroviral therapy (3-6 drugs excluding low-dose ritonavir) for at least 5 months.

Exclusion Criteria:

* Currently receiving maraviroc.
* Active opportunistic infections.
* ALT and/or AST >5x upper limit of normal.
* Direct bilirubin >1.5x upper limit of normal.
* Severe or decompensated liver disease.
* Liver disease unrelated to viral hepatitis infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2011-05-18 (Actual); Primary Completion 2013-04-23 (Actual); Study Completion 2015-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (48):
- United States (24):
  - The Office of Dr. Franco Antonio Felizarta, M.D., Bakersfield, California
  - AIDS Research Alliance, Los Angeles, California
  - Alameda Health System - Highland Hospital, Oakland, California
  - University of California Davis Research, Sacramento, California
  - University of California, Sacramento, California
  - University of California, San Francisco - Hepatitis/HIV Clinical Trials Group (HHCTG), San Francisco, California
  - University of California, San Francisco - Mt. Zion Hospital, San Francisco, California
  - Community AIDS Resource Inc dba Care Resource, Miami, Florida
  - University of South Florida Health - HIV Clinical Research Unit, Tampa, Florida
  - Rowan Tree Medical, P.A., Wilton Manors, Florida
  - Georgia Regents Medical Center, Augusta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Michael's Medical Center, Newark, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Mount Sinai Faculty Practice Associates, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - New York Medical College, Valhalla, New York
  - I.D. Consultants, P.A., Charlotte, North Carolina
  - Kaiser Permanente Sunnybrook Medical Office, Clackamas, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Southwest Infectious Disease Clinical Research Inc., Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University Health Care Center Downtown, San Antonio, Texas
- Fakultni nemocnice Brno, Brno, Czechia
- France (3):
  - Hopital de la Croix Rousse, Lyon
  - Hopital Tenon, Service des Maladies Infectieuses, Paris
  - Centre Hospitalier Cochin Saint Vincent de Paul, Paris
- Germany (6):
  - EPIMED - Gesellschaft fuer epidemiologische und klinische Forschung in der Medizin mbH, Berlin
  - Universitaetsklinikum Bonn, Immunologische Ambulanz HIV, Bonn
  - Klinikum der Universitaet zu Koeln, Cologne
  - ifi - Studien und Projekte GmbH, Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Ludwig-Maximilians-Universitaet, München
- Egyesített Szent István és Szent László Kórház Rendelőintézet, Budapest, Hungary
- Poland (3):
  - EMC Instytut Medyczny S.A. Przychodnia przy ul. Lowieckiej, Wroclaw, Lower Silesian Voivodeship
  - Wojewodzki Szpital Obserwacyjno - Zakazny im. Tadeusza Browicza w Bydgoszczy, Bydgoszcz
  - SPZOZ Wojewodzki Szpital Zakazny, Warsaw
- Puerto Rico (3):
  - Farmacia UPR-CTU, San Juan, PR
  - Ararat Research Center, Ponce
  - University of Puerto Rico - School of Medicine, San Juan
- Spain (5):
  - Hospital Universitari Vall dHebron, Barcelona
  - Hospital Reina Sofia Hospital Provincial, Córdoba
  - Hospital Carlos Iii, Madrid
  - Hospital Nuestra Señora de Valme, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
- United Kingdom (2):
  - Harrison Wing Research Office, Guys and St. Thomas NHS Foundation Trust, London
  - St Stephen's AIDS Trust, London

REFERENCES:
- [Derived] Rockstroh JK, Plonski F, Bansal M, Fatkenheuer G, Small CB, Asmuth DM, Pialoux G, Zhang-Roper R, Wang R, Pineda JA, Heera J. Hepatic safety of maraviroc in patients with HIV-1 and hepatitis C and/or B virus: 144-week results from a randomized, placebo-controlled trial. Antivir Ther. 2017;22(3):263-269. doi: 10.3851/IMP3116. Epub 2016 Dec 7. PMID 27924779
- [Derived] Rockstroh JK, Soriano V, Plonski F, Bansal M, Fatkenheuer G, Small CB, Asmuth DM, Pialoux G, Mukwaya G, Jagannatha S, Heera J, Pineda JA. Hepatic safety in subjects with HIV-1 and hepatitis C and/or B virus: a randomized, double-blind study of maraviroc versus placebo in combination with antiretroviral agents. HIV Clin Trials. 2015 Mar-Apr;16(2):72-80. doi: 10.1179/1528433614Z.0000000011. PMID 25923596
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001098&StudyName=A%20Study%20Of%20Maraviroc%20In%20HIV%20Co-Infected%20Subjects%20With%20Hepatitis%20C%20And/Or%20Hepatitis%20B

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study, 138 participants were randomized, of which 137 participants received the study drug. Participants were randomized at 37 sites in 9 countries. Five sites received drug and screened subjects but did not randomize any subjects; 2 sites received drug but did not screen any subjects.
Pre-assignment Details: One participant who was randomized into the study was withdrawn prior to receiving treatment due to poor venous access.
Groups:
- Maraviroc: Participants who received maraviroc in combination with Highly active antiretroviral therapy (HAART)
- Placebo: Participants who received placebo in combination with HAART
Period: Overall Study
Arm/Group | Maraviroc | Placebo
Started | 70 | 67
Randomized and Not Treated | 0 | 1 (Randomized but was withdrawn prior to receiving treatment due to poor venous access.)
Completed | 50 | 45
Not Completed | 20 | 22
Not completed — Adverse Event | 4 | 1
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 6 | 6
Not completed — Non-Compliance With Study Treatment | 0 | 2
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Does Not Meet Entrance Criteria | 2 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Non-compliance due to alcohol intake | 0 | 1
Not completed — Required prohibited medication | 2 | 0
Not completed — Non-compliance with study procedures | 1 | 0
Not completed — By investigator in subject's interest | 0 | 1

BASELINE CHARACTERISTICS:
Population: A participant was included in the FAS if the participant had taken at least one dose of study drug.
Groups:
- Maraviroc: Participants who received maraviroc in combination with HAART
- Total: Total of all reporting groups
Arm/Group | Maraviroc | Placebo | Total
Number analyzed (Participants) | 70 | 67 | 137
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0
  18-44 years | 26 | 20 | 46
  45-64 years | 42 | 47 | 89
  ≥65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 60 | 57 | 117

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade 3 and Grade 4 Alanine Aminotransferase (ALT) Abnormalities at Week 48
Description: Percentage of participants with Grade 3 or Grade 4 ALT abnormalities defined as >5x upper limit of normal (ULN) for participants whose baseline ALT ≤ULN, or >3.5x baseline for participants whose baseline ALT >ULN, up to and including Week 48 in the maraviroc arm versus the placebo arm. The baseline was defined as the last measurement prior to Day 1 dosing.
Time Frame: 48 weeks
Population: The analysis was performed on the Full Analysis Set (FAS) which included participants who had received at least one dose of study drug. LOCF was used if the value at that time-point was missing, ie., week 48, 96 and 144.
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
Percentage of participants | 1.4 | 1.5
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; A stratified analysis was conducted by summarizing the difference in proportions adjusted for the randomization strata formed by crossing levels of stratification variables. The Cochran-Mantel-Haenszel (CMH) approach was used. No formal hypothesis test was performed; Test type: Superiority or Other; p = 0.4598, Cochran-Mantel-Haenszel; Difference in proportion = -0.0020, 95% CI 2-sided [-0.0417 to 0.0376] — Difference in proportion: CMH approach weighted by hepatitis B virus (HBV) status and usage of protease inhibitor (PI) regimen strata was used to calculate the statistics

2. Secondary Outcome: Percentage of Participants With Grade 3 and Grade 4 ALT Abnormalities Through Week 144
Description: Percentage of participants with Grade 3 or Grade 4 ALT abnormalities defined as >5x upper limit of normal (ULN) for participants whose baseline ALT ≤ULN, or >3.5x baseline for participants whose baseline ALT >ULN, up to and including Week 96 and Week 144 in the maraviroc arm versus the placebo arm. The baseline was defined as the last measurement prior to Day 1 dosing.
Time Frame: Week 96 and 144
Population: The analysis was performed on the FAS which included participant who had received at least one dose of study drug. LOCF was used if the value at that time-point was missing, ie., week 48, 96 and 144.
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
Percentage of participants
  at Week 96 | 1.4 | 3.0
  at Week 144 | 2.9 | 4.5
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.0167, 95% CI 2-sided [-0.0653 to 0.0319] — CMH approach weighted by HBV status and usage of PI regiment strata, is used to calculate the statistics. The point estimate and 95% CI are difference in proportions between MVC and placebo for the participants meeting secondary endpoint
Statistical Analysis 2: Comparison: Maraviroc vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.0177, 95% CI 2-sided [-0.0805 to 0.0452] — CMH approach weighted by HBV status and usage of PI regiment strata, is used to calculate the statistics. The point estimate and 95% CI are difference in proportions between maraviroc and placebo for the participants meeting secondary endpoint

3. Secondary Outcome: Time to Development of Grade 3 and Grade 4 ALT Abnormalities
Description: Time taken in days to development of Grade 3 and Grade 4 ALT abnormalities defined as >5x ULN for participants whose baseline ALT ≤ULN, or >3.5x baseline for participants whose baseline ALT >ULN, at Week 144.
Time Frame: 144 weeks
Population: Time taken in days to development of Grade 3 and Grade 4 ALT abnormalities defined as >5x ULN for participants whose baseline ALT ≤ULN, or >3.5x baseline for participants whose baseline ALT >ULN, at Week 144. The median time to development was not estimable due to too few events reported under each treatment group.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
Days | NA [NA to NA] — Since only 2 participants overall experienced protocol-defined Grade 3 or Grade 4 ALT primary safety endpoint abnormalities during the 48-week period, it was not possible to calculate the median time to primary safety endpoint abnormalities. | NA [NA to NA] — Since only 2 participants overall experienced protocol-defined Grade 3 or Grade 4 ALT primary safety endpoint abnormalities during the 48-week period, it was not possible to calculate the median time to primary safety endpoint abnormalities.

4. Secondary Outcome: Percentage of Participants With Grade 3 and Grade 4 ALT Abnormalities Associated With a Change From Baseline ALT >100 IU/L
Description: Percentage of participants who had Grade 3 and Grade 4 ALT abnormalities associated with a change from baseline ALT >100 IU/L during the 144-week period. Baseline will be defined as the last measurement prior to Day 1 dosing.
Time Frame: 144 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
Percentage of participants
  Grade 3 | 2.8 | 4.4
  Grade 4 | 1.4 | 0.0

5. Secondary Outcome: Time to Development of Grade 3 and Grade 4 ALT Abnormalities at Week 144 Associated With a Change From Baseline ALT >100 IU/L
Description: Time to development of Grade 3 and Grade 4 ALT abnormalities associated with a change from baseline ALT >100 IU/L during the 144-week period. Baseline will be defined as the last measurement prior to Day 1 dosing.
Time Frame: 144 weeks
Population: The analysis was performed on the FAS which included participant who had received at least one dose of study drug. LOCF was used if the value at that time-point was missing, ie., week 48, 96 and 144. The median time to development was not estimable due to too few events reported under each treatment group.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
Days | NA [NA to NA] — Since only 2 participants overall experienced protocol-defined Grade 3 or Grade 4 ALT primary safety endpoint abnormalities during the 48-week period, it was not possible to calculate the median time to primary safety endpoint abnormalities. | NA [NA to NA] — Since only 2 participants overall experienced protocol-defined Grade 3 or Grade 4 ALT primary safety endpoint abnormalities during the 48-week period, it was not possible to calculate the median time to primary safety endpoint abnormalities.

6. Secondary Outcome: Number of Participants With Hy's Law Abnormalities Through Week 144
Description: Hy's law was defined as a total bilirubin >2x ULN with a simultaneous ALT or aspartate transaminase (AST)>3x ULN, excluding participants with an alkaline phosphatase>3x ULN
Time Frame: 144 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
participants | 0 | 0

7. Secondary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) Concentration <40 Copies/mL at Week 48, 96 and 144
Description: The Food and Drug Administration (FDA's) snapshot algorithm was used to derive the efficacy endpoint of the proportion of participants with HIV-1 RNA <40 copies/mL at Week 48. This algorithm included the missing data imputation method and used the plasma HIV-1 RNA concentration in the visit window only, followed the "virology-first principle" and considered a participant who had a missing plasma HIV-1 RNA concentration, or switched to a prohibited background anti-retroviral regimen or discontinues from the study or study drug as a failure (MSDF).
Time Frame: Week 48, 96 and 144
Population: The analysis was performed on the FAS which included participant who had received at least one dose of study drug. For calculating proportions at the analysis timepoint of interest, ie week 144, LOCF was used if the value at that timepoint was missing.
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
Percentage of participants
  Week 48 | 77.1 | 79.1
  Week 96 | 67.1 | 70.1
  Week 144 | 58.6 | 67.2
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; A stratified analysis was conducted by summarizing the difference in proportions adjusted for the randomization strata formed by crossing levels of stratification variables. The CMH approach was used. No formal hypothesis test was performed. Week 48 data presented here; Test type: Superiority or Other; Difference in proportion = -0.0150, 95% CI 2-sided [-0.1484 to 0.1185] — Difference in proportion: CMH approach weighted by HBV status and usage of PI regimen strata was used to calculate the statistics
Statistical Analysis 2: Comparison: Maraviroc vs Placebo; A stratified analysis was conducted by summarizing the difference in proportions adjusted for the randomization strata formed by crossing levels of stratification variables. The CMH approach was used. No formal hypothesis test was performed. Week 96 data presented here; Test type: Superiority or Other; Mean Difference (Final Values) = -0.0255, 95% CI 2-sided [-0.1784 to 0.1274] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Maraviroc vs Placebo; A stratified analysis was conducted by summarizing the difference in proportions adjusted for the randomization strata formed by crossing levels of stratification variables. The CMH approach was used. No formal hypothesis test was performed. Week 144 data presented here; Test type: Superiority or Other; Mean Difference (Final Values) = -0.0830, 95% CI 2-sided [-0.2421 to 0.0761] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Mean Change From Baseline in CD4+ and CD8+ Cell Counts at Week 48, 96 and 144
Description: Immunologic response (magnitude of change in CD4+ and CD8+ cell counts from baseline) was measured. Baseline value for CD4 and CD8 is defined as the pre-dose measurement taken at Day 1 visit.
Time Frame: Week 48, 96 and 144
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Cells/µL
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 69 | 67
Cells/µL
  CD4+ (week 48, n=69, 67) | 3.1 (142.58) | 42.0 (166.35)
  CD8+ (week 48, n=69, 67) | 7.8 (229.53) | 28.9 (293.18)
  CD4+ (week 96, n=69, 67) | 5.1 (146.64) | 49.7 (177.18)
  CD8+ (week 96, n=69, 67) | -2.7 (228.92) | 62.6 (376.67)
  CD4+ (week 144, n=69, 67) | 17.2 (184.86) | 41.7 (200.00)
  CD8+ (week 144, n=69, 67) | 12.6 (293.82) | 44.1 (387.61)
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; The above analysis is for CD4+ cells at week 48. Results are from an analysis of covariance (ANCOVA) model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, hepatitis B virus status (HBV), Protease inhibitor (PI)-based regimen; Test type: Superiority or Other; p = 0.1174, ANCOVA; Difference in Least Square (LS) Mean = -41.12, 95% CI 2-sided [-92.72 to 10.49] — Difference in Least Square (LS) Mean
Statistical Analysis 2: Comparison: Maraviroc vs Placebo; The above analysis is for CD8+ cells at Week 48. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, hepatitis B virus status (HBV), Protease inhibitor (PI)-based regimen; Test type: Superiority or Other; p = 0.5930, ANCOVA; Difference in LS Mean = -21.96, 95% CI 2-sided [-103.05 to 59.12] — Difference in LS Mean
Statistical Analysis 3: Comparison: Maraviroc vs Placebo; The above analysis is for CD4+ cells at Week 96. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, hepatitis B virus status (HBV), Protease inhibitor (PI)-based regimen; Test type: Superiority or Other; p = 0.0669, ANCOVA; Difference in LS Mean = -48.26, 95% CI 2-sided [-99.93 to 3.41]
Statistical Analysis 4: Comparison: Maraviroc vs Placebo; The above analysis is for CD8+ cells at Week 96. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, hepatitis B virus status (HBV), Protease inhibitor (PI)-based regimen; Test type: Superiority or Other; p = 0.1799, ANCOVA; Difference in LS Mean = -65.28, 95% CI 2-sided [-161.07 to 30.50]
Statistical Analysis 5: Comparison: Maraviroc vs Placebo; The above analysis is for CD4+ cells at Week 144. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, hepatitis B virus status (HBV), Protease inhibitor (PI)-based regimen; Test type: Superiority or Other; p = 0.3859, ANCOVA; Difference in LS Mean = -27.71, 95% CI 2-sided [-90.71 to 35.29]
Statistical Analysis 6: Comparison: Maraviroc vs Placebo; The above analysis is for CD8+ cells at Week 144. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, hepatitis B virus status (HBV), Protease inhibitor (PI)-based regimen; Test type: Superiority or Other; p = 0.5571, ANCOVA; Difference in LS Mean = -31.86, 95% CI 2-sided [-138.93 to 75.21]

9. Secondary Outcome: Mean Change From Baseline in CD38 Expression on CD4 and CD8 Cells at Weeks 48, 96 and 144
Description: Plasma samples were used to determine markers of immune activation namely CD38 expression on CD4 and CD8 cells.
Time Frame: 48, 96 and 144 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cell/mm³
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 69 | 67
cell/mm³
  Week 48 (n=69, 67) | -12.2 (129.82) | 43.0 (135.71)
  Week 96 (n=69, 67) | 5.4 (134.64) | 47.4 (186.74)
  Week 144(n=69, 67) | 23.4 (169.50) | 50.7 (219.95)
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; The above analysis is for CD38 expression on CD4 and CD8 cells at Week 48. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.0153, ANCOVA; Difference in LS Mean = -56.06, 95% CI 2-sided [-101.20 to -10.92] — Difference in LS Mean
Statistical Analysis 2: Comparison: Maraviroc vs Placebo; The above analysis is for CD38 expression on CD4 and CD8 cells for Week 96. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.0947, ANCOVA; Difference in LS Mean = -44.93, 95% CI 2-sided [-97.72 to 7.87]
Statistical Analysis 3: Comparison: Maraviroc vs Placebo; The above analysis is for CD38 expression on CD4 and CD8 cells for Week 144. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.3595, ANCOVA; Difference in LS Mean = -29.75, 95% CI 2-sided [-93.74 to 34.24]

10. Secondary Outcome: Mean Change From Baseline in Markers of Immune Activation: C-reactive Protein (CRP) - Week 48, 96 and 144.
Description: Plasma samples were used to determine markers of immune activation namely CRP.
Time Frame: 48, 96 and 144 weeks
Population: The analysis was performed on the FAS which included participants who had received at least one dose of study drug. LOCF was used if the value at that time-point was missing, ie., week 48, 96 and 144.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
mg/dL
  Week 48 (n=70, 67) | 0.4 (8.18) | 3.1 (26.66)
  Week 96 (n=70, 67) | 0.0 (5.16) | -0.7 (3.32)
  Week 144 (n=70, 67) | 0.6 (7.99) | -0.3 (5.28)
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; The above analysis is for C-reactive protein cells at Week 48. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.4476, ANCOVA; Difference in LS Mean = -2.53, 95% CI 2-sided [-9.11 to 4.05] — Difference in LS Mean
Statistical Analysis 2: Comparison: Maraviroc vs Placebo; The above analysis is for C-reactive protein cells at Week 96. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.3012, ANCOVA; Difference in LS Mean = 0.67, 95% CI 2-sided [-0.61 to 1.96]
Statistical Analysis 3: Comparison: Maraviroc vs Placebo; The above analysis is for C-reactive protein cells at Week 144. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.4196, ANCOVA; Difference in LS Mean = 0.92, 95% CI 2-sided [-1.33 to 3.17]

11. Secondary Outcome: Mean Change From Baseline in Markers of Immune Activation: D Dimer - Week 48, 96 and 144
Description: Plasma samples were used to determine markers of immune activation namely D-Dimer.
Time Frame: 48, 96 and 144 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
ng/dL
  Week 48 (n= 68, 65) | -101.1 (753.24) | -20.4 (215.62)
  Week 96 (n= 68, 65) | -88.1 (740.14) | -23.1 (201.55)
  Week 144 (n= 68, 65) | -97.4 (768.98) | 9.8 (358.07)
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; The above analysis is for D-Dimer cells at Week 48. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.9904, ANCOVA — Not specifed; Difference in LS Mean = 0.30, 95% CI 2-sided [-48.66 to 49.26] — Difference in LS Mean
Statistical Analysis 2: Comparison: Maraviroc vs Placebo; The above analysis is for D-Dimer cells at Week 96. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.7697, ANCOVA; Difference in LS Mean = 10.87, 95% CI 2-sided [-62.44 to 84.18] — Difference in LS Mean
Statistical Analysis 3: Comparison: Maraviroc vs Placebo; The above analysis is for D-Dimer cells at Week 144. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.5816, ANCOVA; Difference in LS Mean = -24.49, 95% CI 2-sided [-112.21 to 63.23] — Difference in LS Mean

12. Secondary Outcome: Mean Change From Baseline in Markers of Immune Activation: Transforming Growth Factor-beta (TGF Beta) - Week 48, 96 and 144
Description: Plasma samples were used to determine markers of immune activation namely TGF beta.
Time Frame: 48, 96 and 144 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
ng/L
  Week 48 (n= 67, 66) | 64.1 (4857.31) | -165.0 (2584.89)
  Week 96 (n= 67, 66) | -227.5 (4417.59) | -296.5 (2200.97)
  Week 144 (n= 67, 66) | 792.0 (6772.41) | 1275.4 (5044.79)
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; The above analysis is for TGF-beta cells at Week 48. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.3786, ANCOVA; Difference in LS Mean = 498.04, 95% CI 2-sided [-617.33 to 1613.41] — Difference in LS Mean
Statistical Analysis 2: Comparison: Maraviroc vs Placebo; The above analysis is for TGF-beta cells at Week 96. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.4388, ANCOVA; Difference in LS Mean = 348.70, 95% CI 2-sided [-539.61 to 1237.01] — Difference in LS Mean
Statistical Analysis 3: Comparison: Maraviroc vs Placebo; The above analysis is for TGF-beta cells at Week 144. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.8559, ANCOVA; Difference in LS Mean = -173.57, 95% CI 2-sided [-2060.81 to 1713.68] — Difference in LS Mean

13. Secondary Outcome: Mean Change From Baseline in Log10 Plasma Hepatitis C Virus (HCV) RNA at Week 48, 96 and 144
Description: Plasma samples were used to determine HCV RNA using the Roche COBAS Ampliprep/COBAS HCV Taqman assay, RUO version (LOD=15 IU/mL).Baseline value for HCV RNA/HBV DNA is defined as the pre-dose measurement taken at Day 1 visit.
Time Frame: 48, 96 and 144 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 values
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
Log10 values
  Week 48 (n= 45, 45) | -3.2 (0.60) | -3.2 (0.68)
  Week 96 (n= 45, 45) | -3.2 (0.50) | -3.4 (0.81)
  Week 144 (n= 45, 45) | -3.1 (0.57) | -3.3 (0.72)
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; The above analysis is change for baseline in Log10 plasma HCV RNA at 48 Weeks. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.8024, ANCOVA; Difference in LS Mean = 0.03, 95% CI 2-sided [-0.22 to 0.28] — Difference in LS Mean
Statistical Analysis 2: Comparison: Maraviroc vs Placebo; The above analysis is change for baseline in Log10 plasma HCV RNA at 96 Weeks. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.2660, ANCOVA; Difference in LS Mean = 0.15, 95% CI 2-sided [-0.12 to 0.43] — Difference in LS Mean
Statistical Analysis 3: Comparison: Maraviroc vs Placebo; The above analysis is change for baseline in Log10 plasma HCV RNA at 144 Weeks. Results are from an ANCOVA model with change from baseline as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.2855, ANCOVA; Difference in LS mean = 0.15, 95% CI 2-sided [-0.12 to 0.41] — Difference in LS mean

14. Secondary Outcome: Mean Change From Baseline in Plasma Hepatitis B Virus (HBV) DNA at Week 48, 96 and 144
Description: Plasma samples were used to determine HBV DNA using the Roche COBAS Taqman HBV assay. Baseline value for HCV RNA/HBV DNA is defined as the pre-dose measurement taken at Day 1 visit.
Time Frame: 48, 96 and 144 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 values
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
Log10 values
  Week 48 (n= 15, 10) | -2.6 (1.55) | -3.0 (0.11)
  Week 96 (n= 15, 14) | -3.3 (0.94) | -3.0 (0.00)
  Week 144 (n= 15, 15) | -3.4 (0.96) | -3.0 (0.00)
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; Results are from an ANCOVA model with change from baseline at Week 48 as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.7778, ANCOVA; Difference in LS Mean = 0.15, 95% CI 2-sided [-0.93 to 1.23] — Difference in LS Mean
Statistical Analysis 2: Comparison: Maraviroc vs Placebo; Results are from an ANCOVA model with change from baseline at Week 96 as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.9991, ANCOVA; Difference in LS mean = 0.00, 95% CI 2-sided [-0.10 to 0.10] — Difference in LS Mean
Statistical Analysis 3: Comparison: Maraviroc vs Placebo; Results are from an ANCOVA model with change from baseline at Week 144 as the response variable and the following fixed effect model terms: treatment (Maraviroc or placebo), baseline value of the response variable, HBV, PI-based regimen; Test type: Superiority or Other; p = 0.7275, ANCOVA; Difference in LS mean = -0.02, 95% CI 2-sided [-0.16 to 0.11] — Difference in LS Mean

15. Secondary Outcome: Mean Change From Baseline in Enhanced Liver Fibrosis (ELF) Test at Week 48, 96 and 144
Description: The markers of fibrosis assessed in this test comprised hyaluronic acid (CHA), tissue inhibitor of metalloproteinase (CTIMP1) and procollagen III N-terminal peptide (CP3NP); these are components of the extracellular matrix and basement sinusoidal membrane of the liver and are elevated during activation of the stellate cell. The ELF tests were performed on an ADVIA Centaur XP and the composite score was calculated as follows: ELF score = 2.278 + 0.851 ln(CHA) + 0.751 ln (CP3NP) + 0.394 ln(CTIMP1).
  ELF score < 7.7: no to mild fibrosis; ≥ 7.7 - < 9.8: Moderate fibrosis; ≥ 9.8 - < 11.3: Severe fibrosis; ≥ 11.3: Cirrhosis.
Time Frame: 48, 96 and 144 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ELF score
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
ELF score
  Week 48 (n= 70, 67) | 0.2 (0.70) | 0.1 (0.71)
  Week 96 (n= 70, 67) | 0.4 (0.73) | 0.4 (0.58)
  Week 144 (n= 70, 67) | 0.4 (0.72) | 0.4 (0.69)
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.5201, ANCOVA; Difference in LS Mean = 0.07, 95% CI 2-sided [-0.15 to 0.30] — Difference in LS Mean
Statistical Analysis 2: Comparison: Maraviroc vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.4657, ANCOVA; Difference in LS Mean = -0.08, 95% CI 2-sided [-0.28 to 0.13]
Statistical Analysis 3: Comparison: Maraviroc vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority or Other; p = 0.8087, ANCOVA; Difference in LS Mean = -0.03, 95% CI 2-sided [-0.25 to 0.20] — Difference in LS Mean

16. Secondary Outcome: Mean Change From Baseline in the Hepatic Elastography (FibroscanTM) at Week 48, 96 and 144
Description: Participants had transient hepatic elastography using FibroScan technology. It rapidly and non invasively measures hepatic tissue stiffness. Through a probe, a low frequency vibration of low amplitude is transmitted to the liver. The velocity of the wave that is generated during the procedure correlates directly with tissue stiffness as it passes through the liver; the harder or stiffer the liver, the faster the shear wave propagates. Results are reported in kilopascals (kPa). A negative change in the fibroscan values (i.e. decrease in liver stiffness) correlates with a decrease in fibrosis and thus improved outcome.
Time Frame: 48, 96 and 144 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 25 | 28
kPa
  Week 48 (n= 25, 28) | -1.3 (2.41) | 0.4 (5.71)
  Week 96 (n= 25, 28) | -0.8 (2.95) | 0.4 (5.70)
  Week 144 (n= 25, 28) | -1.7 (2.45) | -0.3 (4.39)
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.1417, ANCOVA; Difference in LS Mean = -1.84, 95% CI 2-sided [-4.31 to 0.63] — Difference in LS Mean
Statistical Analysis 2: Comparison: Maraviroc vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.2679, ANCOVA; Difference in LS Mean = -1.44, 95% CI 2-sided [-4.01 to 1.14] — Difference in LS Mean
Statistical Analysis 3: Comparison: Maraviroc vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority or Other; p = 0.1366, ANCOVA; Difference in LS Mean = -1.48, 95% CI 2-sided [-3.45 to 0.49] — Difference in LS Mean

17. Secondary Outcome: Absolute Fibrosis Score (Ishak) in Liver Biopsy Samples at Baseline and at Week 144
Description: Samples were processed and sent to a central reader for scoring for fibrosis and other analyses such as Sirius red and α smooth muscle actin staining for activated stellate cells. Samples were collected, processed, stored and shipped in accordance with the procedure documented in a separate handling document. The Ishak fibrosis scoring system was used to score the fibrosis observed, with a minimum score of 0 and maximum score of 6 (where 0 = no fibrosis, 1 = expansion of some portal areas with or without septa, 2 = expansion of most portal areas with or without septa, 3 = expansion of most portal areas with occasional portal or portal bridging, 4 = expansion of portal areas with marked bridging [portal-portal and/or portal-central], 5 = marked bridging with occasional nodules [incomplete cirrhosis], 6 = cirrhosis, probable or definitive). The scores for liver biopsies were summarized based upon the availability of liver biopsy results.
Time Frame: Baseline and Week 144
Population: Liver biopsy set consisted of 9 participants (5 MVC and 4 placebo) who had paired baseline and Week 144 liver biopsies that allowed for Ishak fibrosis scoring according to the defined secondary endpoint.
Measure: Mean (Standard Deviation); unit: Numerical score
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 5 | 4
Numerical score
  Absolute Values at Baseline | 2.6 (2.30) [-2.30 to +2.30] | 1.5 (3.0) [-3.0 to +3.0]
  Absolute Values at Post-dose (or Week 144) | 2.2 (1.30) [-1.30 to +1.30] | 1.5 (3.0) [-3.0 to +3.0]

18. Secondary Outcome: Change From Baseline in Fibrosis Score (Ishak) in Liver Biopsy Samples at Week 144
Description: as for outcome 17
Time Frame: Week 144
Population: as for outcome 17
Measure: Median (Full Range); unit: Numerical score
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 5 | 4
Numerical score
  Absolute Values at Baseline | 3 [0 to 6] | 0 [0 to 6]
  Absolute Values at Post-dose (or Week 144) | 2 [1 to 4] | 0 [0 to 6]
  Change from baseline in fibrosis score at Week 144 | 0.0 [-2.0 to 1.0] | 0.0 [0.0 to 0.0]

19. Secondary Outcome: Percentage of Participants Who Were Hospitalized Due to Hepatic Disease Through Week 144
Description: Healthcare resource utilization data was collected using the Healthcare Resource Utilization Questionnaire at all study visits except Screening and Baseline. Other components of healthcare resource utilization, including length of hospital stay, type of ward, associated investigative and therapeutic procedures and concomitant medications were captured from primary and secondary data sources.
Time Frame: 144 Weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 70 | 67
Percentage of participants
  Not Hospitalized | 71.4 | 70.1
  Hospitalized due to Hepatic Disease at least once | 10.0 | 5.0
  Hospitalized, but not due to Hepatic Disease | 95.0 | 95.0

20. Secondary Outcome: Summary of Estimated Maraviroc PK Parameters
Description: Week 4 and Week 48 clinic visits were scheduled such that a trough sample may be taken within a time window of 8-16 hours after the previous dose (Ctrough). Blood samples (4mL) were collected from all participants at the Week 4 and 48 visits.
Time Frame: Week 48
Population: Participants included in the statistical analysis of PK parameters were those receiving maraviroc treatment at Week 48 who had PK data available.
Measure: Median (Full Range); unit: ng/mL
Groups:
- Maraviroc 150 mg: Participants received Maraviroc 150 mg twice a day (BID) in combination with a potent CYP3A4 inhibitor
- Maraviroc 300 mg: Participants received Maraviroc 300mg BID in the absence of a potent CYP3A4 inhibitor and inducer
- Maraviroc 600 mg: Participants received Maraviroc 600 mg BID with a potent CYP3A4 inducer (in absence of inhibitor)
Arm/Group | Maraviroc 150 mg | Maraviroc 300 mg | Maraviroc 600 mg
Number analyzed (Participants) | 31 | 8 | 28
ng/mL
  Cavg | 262 [35 to 455] | 166 [72 to 187] | 309 [79 to 656]
  Cmax | 496 [47 to 768] | 258 [162 to 528] | 915 [133 to 1734]
  Cmin | 127.2 [21.6 to 280.5] | 61.3 [19.5 to 112.9] | 69.2 [17.3 to 250.9]

21. Secondary Outcome: Exposure-response Relationship Between Change From Baseline in Liver Fibrosis Biomarkers Versus MVC Cavg at Week 48
Description: The relationship between change from baseline in liver fibrosis biomarkers (AST, ALT, ALK, BIL, ELF and FSCN) versus MVC Cavg was analyzed using Bayesian methods. P-values were assessed for significance in the relationship between liver fibrosis biomarkers and MVC Cavg. P-value <0.05 was regarded as significantly related.
Time Frame: Week 48
Population: Participants included in the statistical analysis of PK parameters were those receiving maraviroc treatment at Week 48 who had PK and liver fibrosis biomarker data available.
Measure: Number; unit: p-value
Groups:
- Aspartate Transaminase (AST): The p-value of change in AST levels from baseline versus MVC Cavg at Week 48.
- Alanine Transaminase (ALT): The p-value of change in ALT levels from baseline versus MVC Cavg at Week 48.
- Bilirubin (BIL): The p-value of change in BIL from baseline versus MVC Cavg at Week 48.
- Enhanced Liver Fibrosis (ELF): The p-value of change in ELF from baseline versus MVC Cavg at Week 48.
- Fibroscan (FSCN): The p-value of change in FSCN from baseline versus MVC Cavg at Week 48.
- Alkaline Phosphatase (ALK): The p-value of change in ALK from baseline versus MVC Cavg at Week 48.
Arm/Group | Aspartate Transaminase (AST) | Alanine Transaminase (ALT) | Bilirubin (BIL) | Enhanced Liver Fibrosis (ELF) | Fibroscan (FSCN) | Alkaline Phosphatase (ALK)
Number analyzed (Participants) | 67 | 67 | 67 | 67 | 24 | 67
p-value | 0.892 | 0.440 | 0.766 | 0.795 | 0.087 | 0.071

ADVERSE EVENTS:
Time Frame: From the date of signing informed consent form up to 30 days after last dose of the study drug.
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Maraviroc | Placebo
Serious Adverse Events (participants affected / at risk) | 22/70 | 19/67
Other Adverse Events (participants affected / at risk) | 63/70 | 62/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc (N=70) | Placebo (N=67)
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 1
Cataract nuclear (Eye disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia necrotising (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Splenic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Breast calcifications (Reproductive system and breast disorders) | 0 | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Pyschotic disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arthrodesis (Surgical and medical procedures) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc (N=70) | Placebo (N=67)
Angina pectoris (Cardiac disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 3
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Arteriosclerotic retinopathy (Eye disorders) | 1 | 0
Chalazion (Eye disorders) | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 12
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Faecaloma (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 3
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 9
Proctitis (Gastrointestinal disorders) | 0 | 1
Tongue disorder (Gastrointestinal disorders) | 1 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 7
Vomiting (Gastrointestinal disorders) | 5 | 7
Asthenia (General disorders) | 1 | 3
Axillary pain (General disorders) | 0 | 1
Chest pain (General disorders) | 3 | 3
Chills (General disorders) | 1 | 0
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 5 | 3
Feeling abnormal (General disorders) | 1 | 0
Influenza like illness (General disorders) | 3 | 1
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Nodule (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 2 | 3
Pyrexia (General disorders) | 4 | 2
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 3 | 0
Abscess neck (Infections and infestations) | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 1
Acute tonsillitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 10 | 7
Cellulitis (Infections and infestations) | 1 | 1
Chlamydial infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 1
Gastritis viral (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 4 | 1
Gingival abscess (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 3 | 2
Infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 1
Latent tuberculosis (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 9 | 6
Onychomycosis (Infections and infestations) | 1 | 2
Oral candidiasis (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 2 | 1
Oral infection (Infections and infestations) | 1 | 1
Otitis externa (Infections and infestations) | 1 | 2
Otitis media (Infections and infestations) | 3 | 0
Otitis media fungal (Infections and infestations) | 0 | 1
Penile abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 5 | 2
Pneumonia (Infections and infestations) | 0 | 5
Rash pustular (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 4
Rhinitis (Infections and infestations) | 2 | 0
Schistosomiasis (Infections and infestations) | 0 | 1
Secondary syphilis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 5 | 4
Subcutaneous abscess (Infections and infestations) | 2 | 3
Syphilis (Infections and infestations) | 3 | 8
Tinea infection (Infections and infestations) | 1 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 3 | 0
Tooth infection (Infections and infestations) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 11 | 11
Urethritis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 5
Viral infection (Infections and infestations) | 6 | 4
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 2
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 2 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 3
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 1 | 1
Blood pressure increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 3
Transaminases increased (Investigations) | 1 | 0
Viral load increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 10
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 7
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ageusia (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 1
Burning sensation (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Complex regional pain syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 6
Dysaesthesia (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 5
Hypertonia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 3 | 3
Sciatica (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 0 | 2
Abnormal dreams (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 4
Depression (Psychiatric disorders) | 5 | 4
Dissociation (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 5 | 6
Nightmare (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 2
Dysuria (Renal and urinary disorders) | 2 | 2
Haematuria (Renal and urinary disorders) | 0 | 1
Leukocyturia (Renal and urinary disorders) | 1 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 2
Renal cyst (Renal and urinary disorders) | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 1
Pruritus genital (Reproductive system and breast disorders) | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 6
Rash (Skin and subcutaneous tissue disorders) | 5 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 3
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1
Abdominal hernia repair (Surgical and medical procedures) | 0 | 1
Skin lesion excision (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 4 | 3
Hypotension (Vascular disorders) | 1 | 1
Varicose vein (Vascular disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Basedow's disease (Endocrine disorders) | 0 | 1
Hypogonadism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Blepharitis (Eye disorders) | 1 | 0
Eye disorder (Eye disorders) | 1 | 0
Retinopathy hypertensive (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 3
Abdominal symptom (Gastrointestinal disorders) | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Inflammation (General disorders) | 1 | 0
Pain (General disorders) | 2 | 1
Peripheral swelling (General disorders) | 1 | 1
Temperature intolerance (General disorders) | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Body tinea (Infections and infestations) | 0 | 1
Carbuncle (Infections and infestations) | 1 | 0
Chikungunya virus infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 1
Ear infection (Infections and infestations) | 1 | 1
Fungal skin infection (Infections and infestations) | 1 | 1
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Genital herpes simplex (Infections and infestations) | 0 | 1
Gingivitis (Infections and infestations) | 1 | 1
Groin abscess (Infections and infestations) | 0 | 2
Herpes virus infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Mastitis (Infections and infestations) | 1 | 0
Muscle abscess (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Proctitis chlamydial (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 | 0
Amylase increased (Investigations) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 1
Paranoia (Psychiatric disorders) | 0 | 1
Substance abuse (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Urethral discharge (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Genital lesion (Reproductive system and breast disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Prostatic disorder (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Spider naevus (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Menopause (Social circumstances) | 1 | 0
Cataract operation (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Peripheral venous disease (Vascular disorders) | 0 | 1
Endocrine ophthalmopathy (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 0
Epididymitis (Infections and infestations) | 0 | 1
Anal pap smear abnormal (Investigations) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
The median time to development of Grade 3 and 4 ALT abnormalities was not estimable due to too few events reported under each treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.